CLINICAL TRIAL: NCT05363878
Title: Development of a Culturally Grounded, Trauma-Informed Alcohol Intervention With a Reserve-Dwelling First Nation Group
Acronym: NativeHEALTH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34AA028587 (NIH); R34AA028587 (NIH)
Record Dates: First submitted 2022-04-22; First posted 2022-05-06 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Drinking; Trauma, Psychological; Historical Trauma
MeSH Terms: conditions — Alcohol Drinking; Psychological Trauma; Historical Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Native HEALTH Condition (Experimental): Participants randomized to the Native HEALTH condition will complete the Native HEALTH intervention. This is a newly developed cultural program designed to reduce harm from alcohol use and improve quality of life among people in Kingsclear First Nation.
  Interventions: Behavioral: Native HEALTH
- Wait-List Control (No Intervention): Participants randomized to the wait-list control group will complete the Native HEALTH intervention after two months.

INTERVENTIONS:
Behavioral: Native HEALTH — This application proposes the development and initial test of a culturally grounded, trauma informed intervention for alcohol use.
  Other Names: To be named based on community feedback
  Arms: Native HEALTH Condition

SUMMARY:
The objective of this project is to develop and obtain preliminary data on a culturally grounded, trauma-informed alcohol intervention. The specific aims are to (1) use Community-Based Participatory Research methods to deepen partnerships with First Nation through capacity-building and knowledge sharing; (2) collect and apply qualitative data to develop a culturally grounded, trauma-informed alcohol intervention that is focused on historical trauma for use with a First Nation sample; and (3) conduct a pilot RCT study to examine acceptability, sustainability, and initial efficacy data of the intervention compared to waitlist control. This work is important, timely, and innovative. Addressing alcohol use has important implications for the health of Indigenous populations.

DETAILED DESCRIPTION:
Using a Community-Based Participatory Research (CBPR) approach, the investigators will work with community partners to develop a culturally grounded, trauma-informed alcohol intervention. The investigators will collaborate with community partners to design, implement, and evaluate this intervention program. A strength of this approach is that in using existing structures, settings, and resources, this intervention will be able to be more easily sustained over time. This work will occur in two stages. Stage 1a, will occur in two phases; first, talking circles will be used to develop the intervention/manual. In this stage, the investigators will explore their place in the community, identifying important stakeholders, recognizing strengths and resources at the local level, pinpointing settings in the community where research and intervention can potentially or already is taking place, and developing a strong communication and collaboration plan that involves community members and researchers to allow for an exchange of knowledge that is bi-directional. Talking circles will identify Indigenous knowledge and practices related to historical trauma and alcohol use. Benchmark: The end of this first phase will yield a manual. Results from the talking circle will provide important knowledge on the targets, techniques, and mechanisms of change for the intervention, as well as the structure of the intervention, including number and length of sessions, treatment setting, and format (group or individual). Second, the investigators will conduct an open pilot trail that will provide information on the manual, delivery of the intervention, and acceptability of participants. Community members (n = 5) will be recruited to go through the intervention and provide qualitative feedback after each session that will be used to further refine intervention components. Benchmark: Open pilot participants will help further refine the manual for delivery in the randomized pilot trial. During Stage 1b (pilot randomized trial), the investigators will test the feasibility, acceptability, and potential efficacy of the program in a randomized, 2-group pilot clinical trial. Participants (N=60) will be randomized to either a wait-list-control (WLC) group (n=30) or to the culturally grounded, trauma-informed alcohol intervention (n=30). Alcohol outcomes will be assessed at baseline, completion, and 3 and 6 months post-completion. The investigators will evaluate whether the program shows promise relative to the WLC group in terms of alcohol consumption, historical losses and response, well-being, and community connectedness. Benchmarks: Major intermediate objectives are: 1) adequate recruitment volume, 2) achievement of targeted enrollment goals, and 3) follow-up rates >= 85% in Stage 1b pilot trial. In the unlikely scenario that recruitment lags, the investigators will first increase field efforts at flyering and following up recruitment letters. If recruitment continues to lag, the investigators have existing relationships with other Indigenous communities in the nearby area that share the same cultural heritage and language. If follow-up rates lag, telephone follow-ups will be intensified and follow-up incentives will be increased as allowed by budgetary constraints. The investigators will also consider truncating 6-month follow-ups to include only those items necessary for alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Used alcohol in the past week
* Self-identify as a First Nation member
* Reside within the partner community
* Want to cut down or stop alcohol use

Exclusion Criteria:

* Experiencing current psychotic symptoms
* High scores (>10) on the Clinical Institute Withdrawal Assessment for Alcohol, Revised

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-09-29 (Estimated)

PRIMARY OUTCOMES:
Time Line Follow-Back (TLFB) | End of treatment (up to 12 weeks following baseline)
  The TLFB interview will be used to assess alcohol use. The TLFB interview is a calendar-assisted structured interview which provides a way to cue memory so that accurate recall is enhanced. A structured interview of drinking behavior has been found to be the most reliable and valid method of assessing prior alcohol use. The TLFB interview has excellent reliability and validity. It will provide data on the percentage of drinking days, average number of standard drinks consumed per drinking day, drinks consumed per day, and the percentage of heavy drinking days.
Time Line Follow-Back (TLFB) | 3-months post treatment completion
  The TLFB interview will be used to assess alcohol use. The TLFB interview is a calendar-assisted structured interview which provides a way to cue memory so that accurate recall is enhanced. A structured interview of drinking behavior has been found to be the most reliable and valid method of assessing prior alcohol use. The TLFB interview has excellent reliability and validity. It will provide data on the percentage of drinking days, average number of standard drinks consumed per drinking day, drinks consumed per day, and the percentage of heavy drinking days.
Time Line Follow-Back (TLFB) | 6-months post treatment completion
  The TLFB interview will be used to assess alcohol use. The TLFB interview is a calendar-assisted structured interview which provides a way to cue memory so that accurate recall is enhanced. A structured interview of drinking behavior has been found to be the most reliable and valid method of assessing prior alcohol use. The TLFB interview has excellent reliability and validity. It will provide data on the percentage of drinking days, average number of standard drinks consumed per drinking day, drinks consumed per day, and the percentage of heavy drinking days.
Historical Loss and Associated Symptoms Scale | 3-months post treatment completion
  To measure symptoms associated with historical trauma, the Historical Loss Associated Symptoms Scale will be administered. This scales quantify 12 types of symptoms that American Indian people may experience when thinking about historical loss. Participants rate how often they experience each symptom, with response options ranging from 1 (Never) to 5 (Always), such that higher scores indicate more severe historical loss associated symptoms.
Historical Loss and Associated Symptoms Scale | 6-months post treatment completion
  To measure symptoms associated with historical trauma, the Historical Loss Associated Symptoms Scale will be administered. This scales quantify 12 types of symptoms that American Indian people may experience when thinking about historical loss. Participants rate how often they experience each symptom, with response options ranging from 1 (Never) to 5 (Always), such that higher scores indicate more severe historical loss associated symptoms.
Historical Loss and Associated Symptoms Scale | End of treatment (up to 12 weeks following baseline)
  To measure symptoms associated with historical trauma, the Historical Loss Associated Symptoms Scale will be administered. This scales quantify 12 types of symptoms that American Indian people may experience when thinking about historical loss. Participants rate how often they experience each symptom, with response options ranging from 1 (Never) to 5 (Always), such that higher scores indicate more severe historical loss associated symptoms.

SECONDARY OUTCOMES:
Alcohol Use Disorder Identification Test (AUDIT) | End of treatment (up to 12 weeks following baseline)
  The AUDIT is a 10-item self-report instrument designed to identify individuals for whom the use of alcohol places them at risk for alcohol problems or who are experiencing such problems. The AUDIT items ask about the past year, although a few items have no specific time reference. AUDIT total scores can range from 0 to 40, and scores of 8 or above have been used to identify individuals who may be at risk for or who are experiencing alcohol problems. Considerable empirical evidence supports the instrument's internal consistency.
Alcohol Use Disorder Identification Test (AUDIT) | 3-months post treatment completion
  The AUDIT is a 10-item self-report instrument designed to identify individuals for whom the use of alcohol places them at risk for alcohol problems or who are experiencing such problems. The AUDIT items ask about the past year, although a few items have no specific time reference. AUDIT total scores can range from 0 to 40, and scores of 8 or above have been used to identify individuals who may be at risk for or who are experiencing alcohol problems. Considerable empirical evidence supports the instrument's internal consistency.
Alcohol Use Disorder Identification Test (AUDIT) | 6-months post treatment completion
  The AUDIT is a 10-item self-report instrument designed to identify individuals for whom the use of alcohol places them at risk for alcohol problems or who are experiencing such problems. The AUDIT items ask about the past year, although a few items have no specific time reference. AUDIT total scores can range from 0 to 40, and scores of 8 or above have been used to identify individuals who may be at risk for or who are experiencing alcohol problems. Considerable empirical evidence supports the instrument's internal consistency.
Cultural Connectedness Scale | End of treatment (up to 12 weeks following baseline)
  The Cultural Connectedness Scale is a 10-item scale designed to measure three components of cultural connectedness for First Nations individuals: identity, traditions, and spirituality. Participants respond "yes" or "no" to five items assessing whether they engage in cultural practices, rate their agreement with one statement using a 5-point scale ranging from strongly disagree to strongly agree, and rate the frequency of their engagement in cultural activities using four items on a 5-point scale ranging from never to every day. Items are summed to create scale scores ranging from 0 to 25, with higher scores indicating greater cultural connectedness. This scale has been used with adequate reliability.
Cultural Connectedness Scale | 3-months post treatment completion
  The Cultural Connectedness Scale is a 10-item scale designed to measure three components of cultural connectedness for First Nations individuals: identity, traditions, and spirituality. Participants respond "yes" or "no" to five items assessing whether they engage in cultural practices, rate their agreement with one statement using a 5-point scale ranging from strongly disagree to strongly agree, and rate the frequency of their engagement in cultural activities using four items on a 5-point scale ranging from never to every day. Items are summed to create scale scores ranging from 0 to 25, with higher scores indicating greater cultural connectedness. This scale has been used with adequate reliability.
Cultural Connectedness Scale | 6-months post treatment completion
  The Cultural Connectedness Scale is a 10-item scale designed to measure three components of cultural connectedness for First Nations individuals: identity, traditions, and spirituality. Participants respond "yes" or "no" to five items assessing whether they engage in cultural practices, rate their agreement with one statement using a 5-point scale ranging from strongly disagree to strongly agree, and rate the frequency of their engagement in cultural activities using four items on a 5-point scale ranging from never to every day. Items are summed to create scale scores ranging from 0 to 25, with higher scores indicating greater cultural connectedness. This scale has been used with adequate reliability.
Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) | End of treatment (up to 12 weeks following baseline)
  The Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) is a ten-item self-report measure of health-related quality of life. This questionnaire was developed by the NIH to assess five domains: physical function, fatigue, pain, emotional distress, and social health -- all of which are compared relative to United States normative scores. Items are rated on a five-point likert scale.
Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) | 3-months post treatment completion
  The Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) is a ten-item self-report measure of health-related quality of life. This questionnaire was developed by the NIH to assess five domains: physical function, fatigue, pain, emotional distress, and social health -- all of which are compared relative to United States normative scores. Items are rated on a five-point likert scale.
Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) | 6-months post treatment completion
  The Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) is a ten-item self-report measure of health-related quality of life. This questionnaire was developed by the NIH to assess five domains: physical function, fatigue, pain, emotional distress, and social health -- all of which are compared relative to United States normative scores. Items are rated on a five-point likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nichea S Spillane, Ph.D., Principal Investigator — University of Rhode Island; Nicole H Weiss, Ph.D., Principal Investigator — University of Rhode Island
Locations (1):
- Kingsclear First Nation, Fredericton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No